CLINICAL TRIAL: NCT04312191
Title: Using Meditation to Treat Anxiety and Improve Quality of Life in Prostate Cancer Patients Receiving Radiation Therapy
Brief Title: Using Meditation for Oncology Anxiety
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not started and PI is retiring.
Sponsor: Mellar Davis MD (Other)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor-Investigator, Mellar Davis MD, Staff Physician Palliative Care, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0958
Record Dates: First submitted 2020-03-04; First posted 2020-03-18 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Quality of Life; Prostate Cancer; Prostate Cancer Recurrent
Keywords: Meditation with a Mantra; prostate cancer; radiation treatment; anxiety; quality of life; GAD-7; FACT-P
MeSH Terms: conditions — Anxiety Disorders; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to standard of care only (Control Group) versus standard of care plus Meditation with a Mantra (MM) (Test Group) and will be followed for a total of 6 sessions of radiation therapy. Randomization will be executed using a computer-generated schema developed by the study biostatistician and stored in an electronic file.
  The Test Group will be taught MM to use during each radiation treatment session and encouraged to practice MM ad libitum outside of the treatment setting.
  For both the Control and Test Groups, validated questionnaires for anxiety and Quality Of Life will be administered at baseline, Session 3 and Session 6.
  For the Test Group only, a log will be kept by the patient from Session 1 through follow-up, noting the times the MM is practiced. The Test Group will also receive a follow-up phone call on week 10 (one month after Session 6) to record whether the patient has continued to practice MM beyond the study requirements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The Control Group participants (Group A) will be initiating radiation therapy and receiving only standard of care therapy per their Radiation Oncologist.
- Test Group (Experimental): The Test Group participants (Group B) will be initiating radiation therapy and receiving standard of care therapy per their Radiation Oncologist. This group will also be taught mantra-based meditation to use during each radiation treatment session and encouraged to practice MM ad libitum outside of the treatment setting.
  Interventions: Other: Mantra Meditation

INTERVENTIONS:
Other: Mantra Meditation — Mantra-based meditation will be taught using a standard one-word mantra (Om). Om is a non-English word that will help with focus as opposed to an English word which may cause distraction based on the word itself.
  Arms: Test Group

SUMMARY:
The current study is a prospective, interventional, randomized, treatment-controlled study, evaluating the use of Meditation with a Mantra (MM) to decrease anxiety levels and improve Quality of Life (QOL) in prostate cancer patients receiving radiation treatment. The study will be conducted across 6 radiation treatment sessions in men with newly diagnosed prostate cancer, Stage 1 to 3A, and men with recurrent prostate cancer. Patients will receive six radiation sessions with usual care with or without the addition of MM. MM Group patients will be given a log at the beginning of the study to record how long they are meditating and if they found meditation beneficial. The General Anxiety Disorder-7 scale (GAD-7) is a validated tool and will be used to assess anxiety in all participants. The Functional Assessment of Cancer Therapy-Prostate, Version 4 (FACT-P) is a validated measure of QOL in prostate cancer patients and will be used to assess QOL in all participants. A one month follow up phone call will determine if the patients are continuing to use the MM and if they found the practice of MM useful not only in their radiation treatment sessions but in their everyday lives.

DETAILED DESCRIPTION:
The current study is a prospective, interventional, randomized, treatment-controlled study, evaluating the use of MM to decrease anxiety levels and improve Quality of Life (QOL) in prostate cancer patients receiving radiation treatment. The study will be conducted across 6 radiation treatment sessions in men with newly diagnosed prostate cancer, Stage 1 to 3A, and men with recurrent prostate cancer. Approximately forty-six patients will be recruited to allow for forty patients to complete assessments. Twenty-three patients will receive six radiation sessions with MM and will be the Test Group. Twenty-three will receive usual care without MM and will be the Control Group. The Test Group will be taught how to meditate using a standard one-word mantra (Om). The first MM session would be a 30-minute introductory session prior to the first radiation treatment followed by five 20-minute sessions prior to each of the remaining five radiation treatments. The Control Group will receive radiation treatments without MM. During the five 20-minute sessions, the patients will receive a meditation refresher and reinforcement to continue to practice meditation at home. The teaching of MM during all sessions will be done by a dedicated research assistant with a Master of Science in Yoga Therapy. Test Group patients will be given a log at the beginning of the study to record how long they are meditating and if they found meditation beneficial. The General Anxiety Disorder-7 scale (GAD-7) is a validated tool and will be used to assess anxiety in all participants. The Functional Assessment of Cancer Therapy-Prostate, Version 4 (FACT-P) is a validated measure of QOL in prostate cancer patients and will be used to assess QOL in all participants. The GAD-7 and FACT-P will be assessed at baseline, radiation Session 3 and radiation Session 6 to determine the impact of MM on anxiety and QOL, respectively, in the Test Group compared to the Control Group. A one month follow up phone call will determine if the patients are continuing to use the MM and if they found the practice of MM useful not only in their radiation treatment sessions but in their everyday lives.

ELIGIBILITY:
Inclusion Criteria:

1. Males age 18 years and older, at the time of signing the informed consent.
2. Diagnosis of prostate cancer, newly diagnosed or recurrent, scheduled to receive radiation therapy for a minimum of 6 treatments.
3. Participant is willing and able to comply with all protocol requirements and procedures.
4. Capable of giving signed informed consent.

Exclusion Criteria:

1. Current treatment for anxiety with benzodiazepines.
2. Current treatment for generalized anxiety disorder with an Selective Serotonin Reuptake Inhibitor(SSRI) or Serotonin and Norepinephrine Reuptake Inhibitors (SNRI) initiated less than 6 weeks prior to enrollment in the study. Stable therapy for greater than 6 weeks prior to enrollment will be allowed.
3. Current use of meditation treatment or therapy.
4. Significant medical conditions which are likely to result in hospitalization during the study.
5. Any conditions which may interfere with the ability to receive and follow meditation instruction or answer questionnaires.
6. Impaired due to use of drugs or alcohol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 scale (GAD-7) | Change from Baseline GAD-7 at Week 6
  Validated tool to assess anxiety
Functional Assessment of Cancer Therapy-Prostate, Version 4 (FACT-P) | Change from Baseline FACT-P at Week 6
  Validated measure of QOL in prostate cancer patients

SECONDARY OUTCOMES:
Meditation Log | From Session 1 through Session 6 (6 weeks)
  A blank log will be provided for the subjects to record the date and duration of the meditation sessions along with whether the meditation took place on a radiation treatment day and if the subject thought the meditation was helpful.
Telephone Follow-up | four weeks following study completion
  A one month follow up phone call will determine if the patients are continuing to use the MM and if they found the practice of MM useful not only in their radiation treatment sessions but in their everyday lives.

CONTACTS AND LOCATIONS:
Overall Officials: Mellar Davis, MD, Principal Investigator — Geisinger Clinic